CLINICAL TRIAL: NCT01445275
Title: A Comparative Effectiveness Study of Cancer Risk Management for Women at Elevated Genetic Risk of Ovarian Cancer
Brief Title: Cost of Cancer Risk Management in Women at Elevated Genetic Risk for Ovarian Cancer Who Participated on GOG-0199
Status: Withdrawn | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8030; NCI-2011-03467 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-8030; CDR0000712395; GOG-8030 (Other: Gynecologic Oncology Group); GOG-8030 (Other: DCP); GOG-8030 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Fallopian Tube Carcinoma; Hereditary Breast and Ovarian Cancer Syndrome; Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ancillary-Correlative (Health Services Research): Outcome data, such as incidence and stage at diagnosis of ovarian, fallopian tube, and peritoneal cancers; number and timing of screening and serum tests performed; number and timing of pelvic ultrasounds performed; surgical procedures performed; cancer-specific and overall survival (if available); and the incidence, type, and grade of significant adverse events, are collected from the Gynecologic Oncology Group (GOG)-0199 records and analyzed. Cost of each medical intervention is also estimated.
  Interventions: Procedure: Evaluation of Cancer Risk Factors; Other: Medical Chart Review; Other: Study of Socioeconomic and Demographic Variables

INTERVENTIONS:
Procedure: Evaluation of Cancer Risk Factors — Ancillary studies
  Other Names: cancer risk factors evaluation
Other: Medical Chart Review — Ancillary study
  Other Names: Chart Review
Other: Study of Socioeconomic and Demographic Variables — Ancillary studies

SUMMARY:
This research trial collects information about types of treatment and the cost of these procedures in women with elevated genetic risk for ovarian cancer who participated on the Gynecology Oncology Group (GOG)-0199 trial. Gathering information about women at elevated genetic risk for ovarian cancer may help doctors learn more about risk reduction procedures and the cost of these procedures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the cost-effectiveness, defined as cost per quality-adjusted life-year saved, of risk-reducing salpingo-oophorectomy (RRSO) versus ovarian cancer screening (OCS) for women at elevated genetic risk of ovarian cancer over a five-year period, using data from GOG-0199 to model survival.

SECONDARY OBJECTIVES:

I. To estimate the cost-effectiveness, defined as cost per quality-adjusted life-year saved, of RRSO versus OCS for women at elevated genetic risk of ovarian cancer over a lifetime, using stage-specific cohorts and population-based data to model long-term survival. (Exploratory) II. To use value of information (VOI) methodology to set future research priorities aimed at developing evidence-based approaches to the management of women who are at elevated genetic risk of ovarian cancer. (Exploratory)

OUTLINE:

Outcome data, such as incidence and stage at diagnosis of ovarian, fallopian tube, and peritoneal cancers; number and timing of screening and serum tests performed; number and timing of pelvic ultrasounds performed; surgical procedures performed; cancer-specific and overall survival (if available); and the incidence, type, and grade of significant adverse events, are collected from the Gynecologic Oncology Group (GOG)-0199 records and analyzed. Cost of each medical intervention is also estimated.

ELIGIBILITY:
Inclusion Criteria:

* Women who were eligible and evaluable for GOG-0199, a prospective, non-randomized, natural history study
* Data collected from GOG-0199 available

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer who participated in GOG-0199
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01 (Estimated); Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness of RRSO versus OCS | 6 months
  Incidence and stage at diagnosis of ovarian, fallopian tube, and peritoneal cancers in the OCS arm and in the RRSO arm will be collected. This information will be obtained from the CANCER UPDATE FORM (CA-0199) and the Ovarian Surgery Form (C-0199). Summary of the number and timing of screening serum tests, pelvic ultrasound, and surgery procedures will be used to calculate costs, and will be incorporated into the model of Markov stage that corresponds to the study timepoint at which these studies were performed.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States